CLINICAL TRIAL: NCT05033067
Title: The Personal Patient Profile Decision Support for Patients With Bladder Cancer
Acronym: P3BC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of Washington (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Nihal E Mohamed, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-0269; 1R21NR018942-01A1 (NIH)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; shared decision making; behavioral intervention; urinary diversion
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention)
- Intervention (P3-BC) Usual Care (Experimental): intervention + usual care group. In addition to receiving usual care, patients will have access to the aid and related materials before consultation with the physician about cystectomy and urinary diversion.
  Interventions: Behavioral: P3BC

INTERVENTIONS:
Behavioral: P3BC — The decisional aid will be developed to enhance patients' communication about cystectomy and urinary diversions with the clinicians, patients' decisions and preparation for self-care. Program users will be able to choose from a menu to view and print: a) summaries of their responses to inquiry questionnaire about information needed, b) selected statistics about specific side effects and self-care, and c) streamed video vignettes with patient actors of mixed cancer stages, age, sex, and race talking with a clinician about their treatment outcomes and self-care. An automatically printed 2-page output to facilitate discussion will list: 1) decision role preference; 2) the 4 highest ranked information preference sheets; and 3) a summary of personal factors plus suggested discussion topics to address with the clinician. The 2-pages will be provided to the treating physician by the research coordinator before the patient's next consultation appointment.
  Other Names: Personal Patient Profile - Bladder Cancer
  Arms: Intervention (P3-BC) Usual Care

SUMMARY:
There is a pressing need to develop a personalized, value-based decisional tool for bladder cancer patients undergoing radical cystectomy (bladder removal) and urinary diversion to help them with communication with the physicians, shared decision making, and preparation for disease-management and follow-up care. The proposed intervention, the Personal Patient Profile - Bladder Cancer (P3-BC), will be the first intervention to address these issues. Results of this pilot randomized feasibility study will provide evidence of the feasibility and acceptability of the P3-BC and will guide further refinement of the tool for a larger experimental trial, with potential dissemination of the program via the Internet and hand-held computing devices.

ELIGIBILITY:
Inclusion Criteria:

* Patients: cystectomy for MIBC and NMIBC;
* at least 18 years;
* able to communicate in English; and
* competent to give consent.

Exclusion Criteria:

- Existence of other cancers or ongoing cancer treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Acceptability E-scale | Baseline
  Acceptability will be assessed with the six-item Acceptability E-scale. The acceptability is defined as 80% acceptable ratings (using mean score of more than 18 on the scale). Using well-established feasibility criteria to assess: 1) monthly screening rate, 2) monthly enrollment rate, 3) proportion of eligible patients screened who are actually recruited, 4) proportion and demographic and clinical characteristics of patients who decline to participate and reasons for refusal, 5) retention/drop-out rates, and 6) duration and completion rate of study assessments. The AES uses a 5-point response scale for each item (1=not acceptable, 5=highly acceptable). Full score from 0 - 30, with higher score indicating higher overall acceptability
Acceptability E-scale | 1 month followup
  Acceptability will be assessed with the six-item Acceptability E-scale. The acceptability is defined as 80% acceptable ratings (using mean score of more than 18 on the scale). Using well-established feasibility criteria to assess: 1) monthly screening rate, 2) monthly enrollment rate, 3) proportion of eligible patients screened who are actually recruited, 4) proportion and demographic and clinical characteristics of patients who decline to participate and reasons for refusal, 5) retention/drop-out rates, and 6) duration and completion rate of study assessments. The AES uses a 5-point response scale for each item (1=not acceptable, 5=highly acceptable). Full score from 0 - 30, with higher score indicating higher overall acceptability
Acceptability E-scale | 3 month followup
  Acceptability will be assessed with the six-item Acceptability E-scale. The acceptability is defined as 80% acceptable ratings (using mean score of more than 18 on the scale). Using well-established feasibility criteria to assess: 1) monthly screening rate, 2) monthly enrollment rate, 3) proportion of eligible patients screened who are actually recruited, 4) proportion and demographic and clinical characteristics of patients who decline to participate and reasons for refusal, 5) retention/drop-out rates, and 6) duration and completion rate of study assessments. The AES uses a 5-point response scale for each item (1=not acceptable, 5=highly acceptable). Full score from 0 - 30, with higher score indicating higher overall acceptability
Program Evaluation Scale | Baseline
  Investigator-designed 12-items instrument to evaluate participants' opinions and acceptance of study procedures and their satisfaction with the decisional aid. Responses for each item range from strongly agree (1) to strongly disagree (4), with higher scores indicating greater dissatisfaction with the intervention. Full scale ranges from 12-48 with higher scores indicating greater dissatisfaction with the intervention.
Program Evaluation Scale | 1 month
  Investigator-designed 12-items instrument to evaluate participants' opinions and acceptance of study procedures and their satisfaction with the decisional aid. Responses for each item range from strongly agree (1) to strongly disagree (4), with higher scores indicating greater dissatisfaction with the intervention. Full scale ranges from 12-48 with higher scores indicating greater dissatisfaction with the intervention.
Program Evaluation Scale | 3 month followup
  Investigator-designed 12-items instrument to evaluate participants' opinions and acceptance of study procedures and their satisfaction with the decisional aid. Responses for each item range from strongly agree (1) to strongly disagree (4), with higher scores indicating greater dissatisfaction with the intervention. Full scale ranges from 12-48 with higher scores indicating greater dissatisfaction with the intervention.

SECONDARY OUTCOMES:
Shared Decision Making Questionnaire (SDM-Q-9) | Baseline
  Shared decision making will be assessed by the SDMQ-9, a 9-item instrument with full scale from 0-100, higher score indicates more positive attitude towards SDM.
Shared Decision Making Questionnaire (SDM-Q-9) | 1 month
  Shared decision making will be assessed by the SDMQ-9, a 9-item instrument with full scale from 0-100, higher score indicates more positive attitude towards SDM.
Shared Decision Making Questionnaire (SDM-Q-9) | 3 month
  Shared decision making will be assessed by the SDMQ-9, a 9-item instrument with full scale from 0-100, higher score indicates more positive attitude towards SDM.
Decisional Conflict Scale | Baseline
  Consists of 16 item scale measuring effectiveness on decision making. Items are given a score value of 0 = strongly agree, 1 = agree, 2 = neither agree nor disagree, 3= disagree, and 4 = disagree, full scale from 0 - 100 with higher total scores indicating higher decisional conflict.
Decisional Conflict Scale | 1 month
  Consists of 16 item scale measuring effectiveness on decision making. Items are given a score value of 0 = strongly agree, 1 = agree, 2 = neither agree nor disagree, 3= disagree, and 4 = disagree, full scale from 0 - 100 with higher total scores indicating higher decisional conflict.
Decisional Conflict Scale | 3 month
  Consists of 16 item scale measuring effectiveness on decision making. Items are given a score value of 0 = strongly agree, 1 = agree, 2 = neither agree nor disagree, 3= disagree, and 4 = disagree, full scale from 0 - 100 with higher total scores indicating higher decisional conflict.
Brief Symptom Index (BSI-18) | Baseline
  Brief Symptom Index (BSI-18) will be used psychological to assess distress. BSI-18 is a self-report 18-item instrument. Raw scores on the BSI-18 are converted to t-scores based on gender-specific normative data from non-patient community dwelling U.S. adults. A T-score = 50 indicating average function compared to the reference population and a standard deviation of 10, with a higher score indicating more symptom.
Brief Symptom Index (BSI-18) | 1 month
  Brief Symptom Index (BSI-18) will be used psychological to assess distress. BSI-18 is a self-report 18-item instrument. Raw scores on the BSI-18 are converted to t-scores based on gender-specific normative data from non-patient community dwelling U.S. adults. A T-score = 50 indicating average function compared to the reference population and a standard deviation of 10, with a higher score indicating more symptom.
Brief Symptom Index (BSI-18) | 3 month
  Brief Symptom Index (BSI-18) will be used psychological to assess distress. BSI-18 is a self-report 18-item instrument. Raw scores on the BSI-18 are converted to t-scores based on gender-specific normative data from non-patient community dwelling U.S. adults. A T-score = 50 indicating average function compared to the reference population and a standard deviation of 10, with a higher score indicating more symptom.
Control Preferences Scale (CPS) | Baseline
  The Control Preferences Scale (CPS) consists of 5 statements designed to elicit patients' preferences for control over decision making. The CPS involves subjects in making a series of paired comparisons to provide their total preference order over the five statements. Six scores are possible based on the subject's two most preferred roles: active-active, active-collaborative, collaborative-active, collaborative-passive, passive-collaborative, and passive-passive. These scores are grouped as: active (active-active or active-collaborative), collaborative (collaborative-active or collaborative-passive), or passive (passive-collaborative or passive-passive).
The Cancer Rehabilitation Evaluation System Medical Interaction Subscale (CARES-MIS) | Baseline
  The Cancer Rehabilitation Evaluation System (CARES-MIS) - Medical Interaction Subscale will be used to assess perceived problems with communication with providers.
  The CARES - Medical Interaction Subscale includes 11items rated on 5 point scale, where 0 represents "not at all" and 4 represents that problem occurred "very much". Total scores range from 0-44 with higher scores indicating poorer perceived communication.
The Cancer Rehabilitation Evaluation System Medical Interaction Subscale (CARES-MIS) | 1 month
  The Cancer Rehabilitation Evaluation System (CARES-MIS) - Medical Interaction Subscale will be used to assess perceived problems with communication with providers.
  The CARES - Medical Interaction Subscale includes 11items rated on 5 point scale, where 0 represents "not at all" and 4 represents that problem occurred "very much". Total scores range from 0-44 with higher scores indicating poorer perceived communication.
The Cancer Rehabilitation Evaluation System Medical Interaction Subscale (CARES-MIS) | 3 months
  The Cancer Rehabilitation Evaluation System (CARES-MIS) - Medical Interaction Subscale will be used to assess perceived problems with communication with providers.
  The CARES - Medical Interaction Subscale includes 11items rated on 5 point scale, where 0 represents "not at all" and 4 represents that problem occurred "very much". Total scores range from 0-44 with higher scores indicating poorer perceived communication.
Bladder Cancer Knowledge Scale | Baseline
  20 investigator-designed items will evaluate patients' knowledge about bladder cancer.Scores range from 1 (Completely certain that is true) to 5 (Completely certain that is false). Total scale from 20-100, with higher scores indicating less knowledge about bladder cancer.
Bladder Cancer Knowledge Scale | 1 month
  20 investigator-designed items will evaluate patients' knowledge about bladder cancer.Scores range from 1 (Completely certain that is true) to 5 (Completely certain that is false). Total scale from 20-100, with higher scores indicating less knowledge about bladder cancer.
Bladder Cancer Knowledge Scale | 3 months
  20 investigator-designed items will evaluate patients' knowledge about bladder cancer.Scores range from 1 (Completely certain that is true) to 5 (Completely certain that is false). Total scale from 20-100, with higher scores indicating less knowledge about bladder cancer.
Self-Care Difficulty Scale | 1 month
  Self-Care Difficulty Scale - Difficulties in self-care will be assessed through 7 investigator-designed items. Scores range from No (0) or Yes (1), with full scale from 0-7. A higher score indicates greater difficulties in self-care.
Self-Care Difficulty Scale | 3 months
  Self-Care Difficulty Scale - Difficulties in self-care will be assessed through 7 investigator-designed items. Scores range from No (0) or Yes (1), with full scale from 0-7. A higher score indicates greater difficulties in self-care.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Mohamed, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal for individual participant data meta-analysis. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website